CLINICAL TRIAL: NCT03881514
Title: The Effect of Mode of Delivery on Automated Auditory Brainstem Response (AABR) Test
Brief Title: Mode of Delivery on Newborn Hearing Test
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.9.16
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hearing Loss, Neonatal
Keywords: Newborn Hearing Screening; Automated Auditory Brainstem Response; Mode Of Delivery
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neonatal hearing screening may fail due to some perinatal and neonatal factors. It is well known that false positivity increases cost and maternal anxiety and anxiety in the neonatal hearing screening. The effect of the type of delivery to hearing screening is not yet clear. The first automated mode of delivery of babies born in Turkey auditory brainstem response (SAD's), the authors aimed to evaluate the effects of the test results and false positive rate.

newborns were evaluated with brainstem response test. The AABR test was performed before patients were discharged. Perinatal and neonatal variables and AABR test results were recorded retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* records of birth process and
* pregnancy test results of newborns.

Exclusion Criteria:

* newborn;
* She was in a neonatal intensive care,
* congenital / chromosomal anomaly,
* undergoing congenital cmv infection,
* facial / ear deformity,
* families with hearing problems,
* those with hyperbiliromyemia,
* <12 hours after delivery,
* maternal infection,
* dm,
* recurrent abortion,
* smoking,
* plesanta previa,

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients who gave birth in our hospital and who had a hearing test in their newborns will form the study group.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
newborn hearing screening results | 1 week after delivery
  hearing test results of newborns. The test results will be grouped according to the type of birth. The effect of the type of delivery on hearing test results will be investigated. The relationship between vaginal route and cesarean section and hearing test will be the first results.
  hearing test results were evaluated separately for the right and left ear as 'passed the test' and 'left test'.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)